CLINICAL TRIAL: NCT02878148
Title: Conditional Imaging Prescription Strategy as an Alternative to Systematic Unenhanced Computed Tomography for Exploration of Acute Uncomplicated Renal Colic With Lower Radiation Exposure
Brief Title: Conditional Imaging Prescription Strategy for Exploration of Acute Uncomplicated Renal Colic
Acronym: IMAGENCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9656; 2015-A01981-48 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2016-08-19; First posted 2016-08-25 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Acute Renal Colic; Nephrolithiasis
Keywords: Nephrolithiasis; Ureteral stone; Acute renal colic; Ultrasonography; Computed tomography; Diagnosis
MeSH Terms: conditions — Renal Colic; Nephrolithiasis; Ureterolithiasis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with suspected acute uncomplicated renal colic (Experimental): Diagnostic imaging
  Interventions: Device: Diagnostic imaging modalities for suspected renal colic

INTERVENTIONS:
Device: Diagnostic imaging modalities for suspected renal colic — All patients with suspected acute uncomplicated renal colic included will undergo ultrasonography in addition to unenhanced CT of pelvis and abdomen and plain X-ray of the abdomen.
  Imaging examination will be performed according to current guidelines.
  Ultrasonography study and colour doppler will include the kidney, ureterovesical joint and ureters. Unenhanced CT will be performed using a dedicated low-dose protocol.

SUMMARY:
Prospective single centre study aiming at validating a conditional imaging strategy for diagnosis of suspected kidney stone.

Consecutive Emergency department patients referred to the medical imaging department for exploration of a suspected acute uncomplicated renal colic will undergo the following interventions : systematic plain abdominal Xray, systematic ultrasonography and systematic unenhanced CT (with a reduced dose scan), in addition to clinical examination and assessment of body mass index and the Sex, Timing, Origin, Nausea, Erythrocytes (STONE) clinical prediction score for symptomatic stone.

Patients will be followed up at 1 month to record the need for urologic intervention and its type.

The performances of different conditional imaging strategy for the diagnosis of suspected renal colic will be assessed retrospectively. The conditional strategies tested will be based on the patient's stone score and BMI and targeted use of combined plain X-ray and ultrasonography and/or unenhanced CT.

The reference diagnosis for renal colic will be made according to the finding of a ureteral stone or indirect signs of urolithiasis at unenhanced CT.

DETAILED DESCRIPTION:
Plain abdominal Xray, Ultrasonography and unenhanced CT of the abdomen and pelvis will be performed at the time of admission to the imaging department, within 2 days from ED visit and within a 1 hour delay from each other.

Ultrasonography will be interpretated in combination to plain abdominal Xray, and independently from unenhanced CT, by two experienced radiologists blinded to the results of each other.

ELIGIBILITY:
Inclusion criteria:

* Adult patient
* Patient admitted to the Emergency department with suspected acute uncomplicated renal colic

Exclusion criteria:

* Patient presenting with fever (>38°C)
* Patient with persisting pain despite administration of morphinic
* Patient presenting with anuria
* Patients with a single kidney and/or history of chronic renal failure
* Pregnant women or breastfeeding women
* Patient with a history of renal colic
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Diagnostic performances (sensitivity,specificity, calculated according to the tested conditional strategies imaging modality) | Baseline
  Different conditional strategies will be evaluated a posteriori based on the targeted use or not of ultrasonography combined to plain X-ray and/or unenhanced CT, according to the patient's STONE score and BMI.
  The reference diagnosis for renal colic will be made according to the finding of a ureteral stone or indirect signs of urolithiasis at unenhanced CT (gold standard imaging modality)

SECONDARY OUTCOMES:
Radiation exposure dose according to the different imaging strategies tested | Baseline
  The reference strategy will be systematic unenhanced CT.
Diagnostic performances of the tested conditional strategies for the diagnosis of ureteral stone in patients with urethral stone who benefited from urologic management | Baseline
Diagnostic performances of the tested conditional strategies for alternative diagnosis | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Claire FAGET, MD, Principal Investigator — Departement of Medical Imaging - Montpellier University Hospital LAPEYRONIE
Locations (1):
- Departement of Medical Imaging, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided